CLINICAL TRIAL: NCT00487864
Title: In Vivo Confocal Scanning Laser Microscopy of Benign Globular, Homogeneous and Reticular Nevi; Comparison With Dermoscopy and Histopathology
Brief Title: In Vivo Confocal Scanning Laser Microscopy of Benign Nevi
Acronym: CSLM-nevi
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Other Study IDs: 01
Record Dates: First submitted 2007-06-18; First posted 2007-06-19 (Estimated); Last update posted 2007-06-19 (Estimated); Status verified 2007-06

CONDITIONS: Nevus
MeSH Terms: conditions — Nevus

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
In vivo confocal laser scanning microscopy (CLSM) offers the possibility to non-invasively investigate skin lesions at nearly histologic resolution. A recent study showed a high sensitivity (97.6%) and specificity (88.15%) for the discrimination of clinical clear cut melanocytic lesions. CSLM provides horizontal images and can be seen as missing link between dermoscopy and histopathology. For a more accurate diagnosis of dermoscopically difficult to diagnose melanocytic skin lesions in the grey zone between nevus and melanoma, the knowledge of CLSM features of benign nevi seems to be essential. We investigated 30 flat benign nevi with different dermoscopic patterns (10 reticular, 10 globular, 10 homogeneous) nevi. CLSM images were assessed in terms of cytomorphologic and architectural criteria. Different dermoscopic patterns of benign nevi are reflected in different architectural features in CLSM.

DETAILED DESCRIPTION:
This study included 29 patients, which were recruited consecutively at our pigmented skin lesion clinic at the Department of Dermatology, University Hospital Graz, Austria. A total of 30 benign nevi were imaged; 10 dermoscopically reticular, 10 globular and 10 homogeneous nevi were selected. Lesions were selected for the presence of a uniform dermoscopic pattern. A biopsy of one nevus of each group was performed due to cosmetic purposes on patient's request.

Each nevus was imaged with a confocal scanning laser microscope (Vivascope 1000, Lucid Inc, Henrietta, NY). Technical details of the confocal scanning microscope have been described elsewhere. The adaptor ring of the laser microscope was applied to the skin and centered on the lesion. A standardized evaluation was performed; CSLM imaging of the lesion centre was started stepwise (approximately 20µm per step) beginning from stratum corneum to the papillary dermis with a field of view of 475 x 350 µm for a single image (´stack´ image). Each image corresponds to a horizontal section at a selected depth with a resolution of 640x480 pixels and 255 colors (grey scale). An automated stepper was used to obtain a grid of 16 contiguous horizontal images of the basal layer, constructing a montage image with a 1.9x1.4mm field of view (´block´ image). Since selected nevi showed a uniform pigmentation pattern throughout the whole lesion, a correlation between clinical, dermoscopic and confocal images could be guaranteed. One nevus of each group was consecutively biopsied and assessed with conventional histopathologic examination after sectioning and staining with hematoxylin and eosin (H&E).

Cytomorphologic and architectural features of each nevus were evaluated during assessment of confocal images and distinct characteristics for each group of nevi were determined and correlated with dermoscopy and, if available, with histopathology. The diagnostic applicability of CSLM in the differentiation between reticular, globular and homogeneous nevi based on these features was assessed by two independent observers.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a benign, flat, dermoscopically uniform pigmented nevus.

Exclusion Criteria:

* Absence of a benign, flat, dermoscopically uniform pigmented nevus.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-09; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Hofmann-Wellenhof, Prof., Principal Investigator — Department of Dermatology, Medical University Graz, Austria
Locations (1):
- Department of Dermatology and Venerology, University Hospital Graz, Graz, Styria, Austria